CLINICAL TRIAL: NCT04820712
Title: Surgical Therapy and Survival in Young Patients With Stage I-II Hepatocellular Carcinoma: A Retrospective Cohort Study
Brief Title: Surgical Therapy and Survival in HCC/ C.F. Zhang et al.
Status: Completed | Type: Observational
Sponsor: Linzhu Zhai (Other)
Responsible Party: Sponsor-Investigator, Linzhu Zhai, Director, The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine
Organization: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other)
Other Study IDs: FirstAHGTCMU
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Hepatocellular Carcinoma; Surgery
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study utilizes a new method to explore compare the overall survival (OS) and cancer-specific survival (CSS) in patients aged 18-45 years with stage I-II HCC who underwent different types of surgery. The SEER database, which is one of the most comprehensive and authoritative databases concerning cancer, was used to estimate the survival benefit of patients who underwent local tumor destruction (LTD), wedge or segmental resection (WSR), lobectomy resection (LR), liver transplantation (LT), or non-surgery. This study discovered surgery offered a survival benefit compared with non-surgery for young patients with stage I-II HCC. Furtherly, LT is associated with superior survival than WSR, LR and LTD in those patients. Our results facilitate the selection of surgical strategies.

DETAILED DESCRIPTION:
The SEER data contain no identifiers and are publicly available for studies of cancer-based epidemiology and survival analysis. Therefore, the current study was deemed to be exempt from Institutional Review Board approval and the need for informed consent was waived. The submitted magazine requires registration on the website, so this operation is needed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were diagnosed with colorectal cancer only;
2. Patients with simultaneous metastasis of liver and lung cancer cells;
3. Patients without metastasis resection;
4. whether they underwent palliative primary tumor resection was known;
5. Their cause of death was known;
6. Their survival time were known and greater than 0 month;
7. Patients were diagnosed with microscopic confirmation.

Exclusion Criteria:

* No

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients aged 18-45, regardless of race。
Sampling Method: Non-Probability Sample
Enrollment: 664 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2004.1.1-2013.12.31
  Overall survival was defined as the duration between the surgery and death or the last follow-up

SECONDARY OUTCOMES:
Cancer-specific survival | 2004.1.1-2013.12.31
  Cancer-specific survival was defined as the period between the surgery and death due to cancer to reduce the impact of life-threatening comorbidities.

CONTACTS AND LOCATIONS:
Locations (1):
- linzhu Zhai, Guangzhou, Guangdong, China

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT04820712/Prot_SAP_ICF_000.pdf